CLINICAL TRIAL: NCT06780462
Title: Randomized Controlled Multicenter Study Comparing Steroid Therapy Plus Anticoagulants to Steroid Therapy Alone in Deep Venous Thrombosis of Behçet's Syndrome
Acronym: ACTOR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP220673
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — Adrenal Cortex Hormones; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, multicentre, superiority study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroids and Rivaroxaban (Experimental)
  Interventions: Drug: Corticosteroids + Rivaroxaban
- Corticosteroids alone (Active Comparator)
  Interventions: Drug: Corticosteroids alone

INTERVENTIONS:
Drug: Corticosteroids + Rivaroxaban — Corticosteroids according to the schedule of reduction of prednisone (or equivalent prednisone dose only if prednisone is out of stock in the market) and Rivaroxaban
  Arms: Corticosteroids and Rivaroxaban
Drug: Corticosteroids alone — Corticosteroids according to the schedule of reduction of prednisone (or equivalent prednisone dose only if prednisone is out of stock in the market)
  Arms: Corticosteroids alone

SUMMARY:
In patients with Behçet's syndrome (BS), deep venous thrombosis (DVT) is thought to result from inflammation of the vessel wall rather than hyper coagulability.

Post Thrombotic Syndrome (PTS) is frequent especially with recurrent episodes of deep vein thrombosis and may result in leg ulcers that are very difficult to treat. Vascular involvement is a major cause of morbidity and mortality among BS patients. However, one of the most controversial issues regarding the management of BS is whether DVT should be treated with anticoagulants. Moreover, use of anticoagulants exposes patients to serious bleeding, especially in those who presents simultaneous arterial aneurysms. However, many physicians are still using anticoagulants. This is the first prospective, randomized study assessing benefits of corticosteroids associated with anticoagulant compared to that of corticosteroids alone in DVT in BS patients. It will validate or not the use of anticoagulants in those situations. It will allow a direct comparison of the safety profile of those two schemes of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Diagnosis of BS according to the international criteria
3. First or recurrent deep venous thrombosis diagnosed on imaging (venous ultrasonography , and/or Angio CT scan and/or angio MRI)
4. Written inform consent
5. Women of childbearing potential (WOCBP) are required to have a negative pregnancy test before treatment and must agree to maintain during treatment highly effective contraception (ie, abstinence, combined estrogen- and progestogen- containing hormonal contraception, ovulation inhibitors (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner).
6. Affiliation to a social security system. Patients affiliated to universal medical coverage (CMU) are eligible for the study

Exclusion Criteria:

1. Clinical condition, other than venous thrombosis, requiring anticoagulation (e.g. atrial fibrillation…)
2. Active bleeding or high risk for bleeding contraindicating treatment with anticoagulants
3. Isolated superficial thrombosis without concomitant deep venous thrombosis.
4. Pregnancy or lactation
5. Have been taking an oral daily dose of a glucocorticoid of more than 20 mg prednisone equivalent for more than 6 weeks continuously prior to the inclusion visit or taking more than 4000 mg methylprednisolone 4 weeks prior to the inclusion visit
6. Have been taking anti-coagulation therapy for more than 4 weeks prior to inclusion
7. Severe chronic renal (creatinine clearance <30ml/min/1,73m2) or liver insufficiency associated with coagulopathy
8. Platelet count < 50 x 103/mm3
9. Change in the treatment with systemic biologic therapy or immunosuppressant therapy dose 1 month prior to inclusion visit.
10. Contraindication to investigational medicinal products (Corticosteroids and direct oral anticoagulant (Rivaroxaban))
11. Participation to another interventional clinical trial or being in the exclusion period at the end of a previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Rate of success | At 6 months
  Defined as absence of deep venous thrombosis relapse and of major bleeding event, without introduction of additional immunosuppressive medication for BS activity other than thrombotic events at 6 months.

SECONDARY OUTCOMES:
Cumulative incidence of deep venous thrombosis and superficial venous thrombosis relapse | At 12 months
Cumulative incidence of major venous thrombosis | At 12 months
  pulmonary embolism, vena cava , Budd Chiari syndrome , intra-cardiac relapse
Cumulative incidence of venous repermeabilization | At 6 months
  assessed by vascular imaging
Proportion of patients with a dose ≤ 5 mg/day of prednisone | At 6 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Proportion of patients with a dose ≤ 5 mg/day of prednisone | At 12 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Dose of prednisone | At 3 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Dose of prednisone | At 6 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Dose of prednisone | At 12 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Cumulative dose of prednisone | At 3 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Cumulative dose of prednisone | At 6 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Cumulative dose of prednisone | At 12 months
  (prednisone or equivalent prednisone dose only if prednisone is out of stock in the market)
Cumulative incidence of major bleeding event | At 12 months
Cumulative incidence of bleeding event | At 12 months
Number of adverse events | At 3 months
Number of adverse events | At 6 months
Number of adverse events | At 12 months
Change in SF-36 quality-of-life | At 3 months
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
Change in SF-36 quality-of-life | At 6 months
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
Change in SF-36 quality-of-life | At 12 months
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
Change in Behçet's Disease Current Activity Form | At 3 months
  It is a 7 items score ranging from 0 to 12. The higher the sore the higher the severity of the disease.
Change in Behçet's Disease Current Activity Form | At 6 months
  It is a 7 items score ranging from 0 to 12. The higher the sore the higher the severity of the disease.
Change in Behçet's Disease Current Activity Form | At 12 months
  It is a 7 items score ranging from 0 to 12. The higher the sore the higher the severity of the disease.
Change in Behçet's Syndrome Assessment Score | At 3 months
  It is based on various clinical manifestations of Behçet's disease. Score ranges from 0 to 12. The higher the score the higher the severity of the disease.
Change in Behçet's Syndrome Assessment Score | At 6 months
  It is based on various clinical manifestations of Behçet's disease. Score ranges from 0 to 12. The higher the score the higher the severity of the disease.
Change in Behçet's Syndrome Assessment Score | At 12 months
  It is based on various clinical manifestations of Behçet's disease. Score ranges from 0 to 12. The higher the score the higher the severity of the disease.
Change in Physician Global Assessment | At 3 months
  Evaluation of the disease activity. It ranges from 0 to 10. The higher the score the higher the activity of the disease.
Change in Physician Global Assessment | At 6 months
  Evaluation of the disease activity. It ranges from 0 to 10. The higher the score the higher the activity of the disease.
Change in Physician Global Assessment | At 12 months
  Evaluation of the disease activity. It ranges from 0 to 10. The higher the score the higher the activity of the disease.
Overall survival | At 12 months
Event free survival | At 12 months
Proportion of post thrombotic syndrome | At 12 months
  According to Villalta's post-thrombotic syndrome scale. It assesses the prensece and severity of post thrombotic syndrome. The score ranges from 0 to 30. The higher the score the more severe are the symptoms
Changes in Villalta's post-thrombotic syndrome scale | At 6 months
  According to Villalta's post-thrombotic syndrome scale. It assesses the prensece and severity of post thrombotic syndrome. The score ranges from 0 to 30. The higher the score the more severe are the symptoms
Changes in Villalta's post-thrombotic syndrome scale | At 12 months
  According to Villalta's post-thrombotic syndrome scale. It assesses the prensece and severity of post thrombotic syndrome. The score ranges from 0 to 30. The higher the score the more severe are the symptoms
Proportion of remission | At 3 months
  According to other organs involved
Proportion of remission | At 6 months
  According to other organs involved
Proportion of remission | At 12 months
  According to other organs involved
Changes in acute-phase reactants | At 1 month
Changes in acute-phase reactants | At 3 months
Changes in acute-phase reactants | At 6 months
Changes in acute-phase reactants | At 12 months

IPD SHARING:
Plan to Share IPD: Undecided